CLINICAL TRIAL: NCT01056393
Title: Investigator-Sponsored Protocol - Continued Use of Ibalizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: TaiMed Biologics Inc. (Industry)
Responsible Party: Principal Investigator, William J. Towner, Partner Physician, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5460
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — ibalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ibalizumab 800mg Q2Weeks (Experimental): Subject will receive 800mg of ibalizumab every 2 weeks administered by intravenous infusion. All patients also will receive optimized background regimen
  Interventions: Drug: ibalizumab 800mg Q2Weeks
- ibalizumab 2000mg Q4Weeks (Experimental): Subject will receive 2000mg of ibalizumab every 4 weeks administered by intravenous infusion. All patients also will receive optimized background regimen
  Interventions: Drug: ibalizumab 2000mg Q4Weeks

INTERVENTIONS:
Drug: ibalizumab 800mg Q2Weeks — Ibalizumab is a humanized IgG4 monoclonal antibody and is provided as a parenteral formulation at a concentration of 25mg/mL in a 10mL glass vial, 8mLs per vial, as the investigational product. Study drug will be administered via intravenous infusion at doses of 800mg every 2 weeks.
  Other Names: TNX-355; TMB-355
  Arms: ibalizumab 800mg Q2Weeks
Drug: ibalizumab 2000mg Q4Weeks — Ibalizumab is a humanized IgG4 monoclonal antibody and is provided as a parenteral formulation at a concentration of 25mg/mL in a 10mL glass vial, 8mLs per vial, as the investigational product. Study drug will be administered via intravenous infusion at doses of 2000mg every 4 weeks.
  Other Names: TNX-355; TMB-355
  Arms: ibalizumab 2000mg Q4Weeks

SUMMARY:
This protocol serves to extend the successful treatment for HIV positive patients beyond the endpoints provided by the Phase 2b TaiMed Biologics-sponsored protocol TMB202 (entitled "A Phase 2b Randomized, Double-Blinded, 48-Week, Multicenter, Dose-Response Study of Ibalizumab Plus an Optimized Background Regimen in Treatment-Experienced Patients Infected with HIV-1 (Amended to 24 Week Study)"), for 24 weeks. Ibalizumab may be administered beyond 24 weeks under this protocol as supply permits and patients continue to demonstrate virologic response.

DETAILED DESCRIPTION:
Ibalizumab is to be administered to HIV-infected patients that have responded (defined as a minimum 0.7 log10 decline in HIV-1 viral load from TMB-202 Baseline) on the TMB-202 protocol. In addition to the investigator-selected Optimized Background Regimen, patient(s) will continue to receive the TMB-202 randomized dose of ibalizumab in open-labeled fashion (800mg IV every two weeks or 2000mg IV every four weeks) as per their original drug assignment for the TMB-202 protocol.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and have voluntarily signed the ICF
* Have documented HIV-1 infection
* Have successfully completed Protocol TMB202 (Amendment 2)(Week 16)
* Have had at least a 0.7 log10 decline in HIV-1 RNA from baseline at Week 16 and beyond while in TMB202 and are no longer eligible to participate in TMB-202 due to TMB-202 protocol-defined virologic failure
* Have not withdrawn or been discontinued from TMB202 9Amendment 2) for any reason
* Are able and willing to comply with all protocol requirements and procedures
* Are 18 years of age or older
* If sexually active, are willing to use an effective method of contraception during the study and for 30days after the last administration of the study drug.

Exclusion Criteria:

* Any active AIDS-defining illness per Category C except for cutaneous Kaposi's sarcoma and wasting due to HIV
* Any significant disease (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, medical history and/or physical examination that, in the investigator's opinion, would preclude the patient from participating in this study
* Any current alcohol or illicit drug use that, in the investigator's opinion, will interfere with the patient's ability to comply with the study schedule and protocol evaluations
* Any previous clinically significant allergy or hypersensitivity to any excipient in the ibalizumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Laboratory testing that includes routine HIV-1 viral load and CD4+ cell counts will be completed to assess the continued benefit of ibalizumab to the patient's HIV treatment. | Every two months

CONTACTS AND LOCATIONS:
Overall Officials: William Towner, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Southern California, Los Angeles, California, United States